CLINICAL TRIAL: NCT07252245
Title: Pre Hospital Triage of Patients at Intermediate and High Risk for ACS: ARTICA-2 Trial
Brief Title: Pre Hospital Triage of Patients at Intermediate and High Risk for ACS
Acronym: ARTICA-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cyril Camaro (Other)
Collaborators: Ambulance services Veiligheidsregio Gelderland-Zuid (Unknown); Canisius Wilhelmina Ziekenhuis (CWZ) (Unknown); Slingeland Hospital (Other); Maas Hospital Pantein (Other); Rijnstate Hospital (Other); RAV Brabant MWN (Other)
Responsible Party: Sponsor-Investigator, Cyril Camaro, Cyril Camaro, PI ARTICA-2, Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL-010807; 10390042410064 (Other: ZonMw - The Netherlands Organisation for Health Research and Development)
Record Dates: First submitted 2025-09-30; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome
Keywords: HEART score; NSTE-ACS; Pre-hospital triage; high risk ACS; intermediate risk ACS; point-of-care troponin

STUDY DESIGN:
Intervention Model Description: Strategy study:
  A) intervention group: Integrating the HEAR score and hs POC troponin: pre- hospital triage decision-making for intermediate and high risk patients:
  B) Standard care group: all intermediate and high risk patients are referred to the nearest hospital to rule-out or rule-in ACS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Integrating the HEAR score and hs POC troponin into pre hospital triage decision-making:
  Interventions: Other: Integrating the HEAR score and hs POC troponin into pre hospital triage decision-making:
- Standard care group (No Intervention): intermediate and high risk patients referred to the nearest hospital for standard care. The ACS rule-out protocol follows the 2023 Guidelines of the European Society of Cardiology (ESC). In confirmed cases of ACS, patients should be scheduled for invasive coronary angiography within the recommended time window as outlined by the ESC guidelines

INTERVENTIONS:
Other: Integrating the HEAR score and hs POC troponin into pre hospital triage decision-making: — Integrating the HEAR score and hs POC troponin into pre hospital triage decision-making: low risk (HEAR score 4 and hs POC troponin < 99th percentile upper reference limit (URL)) will be treated conservatively (i.e. referred to the general practitioner); intermediate risk (HEAR score ≥5 and hs POC troponin < 99th percentile URL or HEAR score 4-6 with intermediate elevated hs POC troponin (i.e. hs POC troponin between 1 and 3 times the 99th percentile URL) are admitted to the nearest hospital with a rapid rule out strategy or recommendation for fast-track coronary CT imaging (CTCA); high risk group (HEAR ≥ 7 ánd hs POC troponin > 99th percentile URL or any HEAR score with hs POC troponin 3x > 99th URL will be directly referred to a PCI center
  Arms: Intervention group

SUMMARY:
RESEARCH QUESTION: Is a treatment strategy that includes direct referral to a PCI center for intermediate to high-risk patients with non-ST elevation acute coronary syndrome (NSTE-ACS), both cost-effective and non-inferior for major adverse cardiac events (MACE)? HYPOTHESIS: Prehospital triage with the modified [History-ECG-Age-Risk factors] (HEAR) score and a high sensitivity (hs) point-of-care troponin (POCT) leads to a faster diagnosis of ACS, faster time to coronary angiography (CAG) and/or treatment with PCI, shorter length of stay, quicker availability of ambulances and more satisfaction and quality of life of patients. STUDY DESIGN: Randomized clinical trial. STUDY POPULATION: Patients ≥18 years with an intermediate to high risk for NSTE -ACS (defined as a modified HEAR score ≥ 4) INTERVENTION: applying modified HEAR score and hs POCT to identify patients for direct rule out (very low risk), transfer to the nearest hospital for rapid rule-out and/or fast-track diagnosis by CT coronary imaging (intermediate risk) or direct referral to a PCI center for CAG (high risk).

USUAL CARE/COMPARISON: Assessment of ACS at the nearest hospital. In case PCI is scheduled: transfer to nearest PCI center.

OUTCOME MEASURES: primary endpoints: healthcare costs and non-inferiority for MACE (all cause death, confirmed ACS, re ACS, and unplanned PCI or CABG) at 30 days. Secondary: MACE after rule out ACS at 30 days, Quality of life (EQ5D5L) and cost-effectiveness at 12 months.

SAMPLE SIZE: 1048 patients. COST-EFFECTIVENESS ANALYSIS / BIA: It is expected that the intervention group will reduce healthcare costs and potentially improve health-related quality of life in this target population. Cost-effectiveness will be expressed as cost per QALY gained. We assume a large potential saving more than € 37 million if 100% implemented. TIME SCHEDULE: 48 months; 36 month inclusion, follow-up 12 months

DETAILED DESCRIPTION:
Rationale: Each year, 230.000 patients in the Netherlands seek medical attention for acute chest pain. The majority of these patients (67%) are at intermediate to high risk of developing non-ST elevation acute coronary syndrome (NSTE-ACS). Immediate ambulance transport to the nearest emergency department (ED) remains the standard of care. The availability of clinical decision rules, along with new high-sensitivity (hs) POC troponin analyzers, presents new opportunities for the early identification of higher-risk patients, potentially improving healthcare logistic. Currently, only observational data are available regarding these groups. Randomized clinical trials (RCT) on a prehospital strategy that includes a rapid rule out or fast-track diagnosis care path for the intermediate risk group or direct referral to a PCI center for the higher risk group has not been studied in a RCT before. More data are needed on prehospital strategies in high-risk groups, focusing on costs and major adverse cardiac events (MACE).

Objective: To assess healthcare costs and safety (MACE) at 30 days of an integrated pre-hospital triage strategy using the [History-ECG-Age-Risk factors] HEAR score and hs POC troponin for patients at intermediate to high risk of NSTE ACS. Secondary objective includes MACE after rule-out ACS at 30 days and cost-effectiveness and quality of life at 12 months.

Study design: Randomized clinical trial (pragmatic strategy trial) Sample size calculation: 1048 patients. A MACE rate of 20% for all risk groups in both the standard and intervention groups: sample sizes of 476 per group to achieve 80% power to detect a non-inferiority margin of 0.0800. The reference group proportion is 0.2000, and the treatment group proportion is 0.2800 under the null hypothesis of inferiority. Power was calculated assuming the actual treatment group proportion is 0.2 Study population: Patients ≥18 years with an intermediate to high risk for NSTE-ACS (defined as a modified HEAR score ≥ 4) Intervention: applying modified HEAR score and hs POC troponin to identify patients for direct rule out (low risk), transfer to the nearest hospital for rapid rule-out and/or fast-track diagnosis in which non-invasive imaging is strongly recommended (intermediate risk) or direct referral to a PCI center (high risk).

Main study parameters/endpoints: primary endpoints: healthcare costs and non-inferiority for MACE (all cause death, confirmed ACS, re ACS, and unplanned PCI or CABG) at 30 days. Secondary: MACE after ruling out ACS at 30 days, Quality of life (EQ5D5L) and cost-effectiveness at 12 months.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Two-thirds of ACS patients are intermediate to high risk and standard hospital evaluation remain the standard of care. In this study the randomized group will receive a patient tailored prehospital management (conservative, local hospital with non-invasive imaging testing, or direct PCI referral). This strategy may safely reduce unnecessary hospitalizations, costs and efficient hospital transfers. While increasing the time to diagnosis of NSTE ACS

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* All out-of-hospital patients with chest pain or symptoms suggestive of ACS with an indication for transfer to the (cardiac) emergency department to evaluate and rule out ACS
* Modified HEAR(T) score ≥ 4
* The patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

* Electrocardiographic ST-segment elevation (STEMI)
* Patients with confirmed myocardial infarction, PCI or CABG <14 days prior to inclu-sion
* Patients presenting an obvious non-cardiac cause for the chest complaints who need evaluation at an emergency department, e.g. trauma, pneumothorax, sepsis, etc.
* Patients in comatose state, defined as an EMV <8
* Patients with known cognitive impairment
* Pregnancy or intention to become pregnant during the course of the study
* Patients presenting with cardiogenic shock, defined as: systolic blood pressure <90mmHg and heart rate >100 and peripheral oxygen saturation <90% (without oxygen administration)
* Patients presenting with syncope
* Patients presenting with signs of heart failure
* Patients presenting with second or third degree atrioventricular block
* Patients without known supraventricular tachycardia i.e. unknown atrial fibrillation (known atrial fibrillation with adequate rate control can be included)
* Patients with known end-stage renal disease (dialysis and/or GFR < 30 ml/min)
* Patients without a pre-hospital 12-lead ECG performed or available
* Patients suspicious of aortic dissection or pulmonary embolism
* Communication issues with patient/language barrier
* Any significant medical or mental condition, which in the Investigator's opinion may interfere with the patient's optimal participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1048 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority for MACE | from enrollment to end of treatment at 30 days and 12 months
  MACE (% all cause death, confirmed ACS, re ACS, and unplanned PCI or CABG). Risk differences will be calculated along with 95% confidence intervals
Healthcare costs | from enrollment to end of treatment at 30 days and 12 months
  healthcare costs in EURO

SECONDARY OUTCOMES:
MACE after ruling out ACS | from enrollment to end of treatment at 30 days
  30-day incidence of MACE in %. Risk differences will be calculated along with 95% confidence intervals
Quality of life measured with the EQ5D5L | from enrollment to end of treatment at 30 days and 12 months
  Quality of life
Cost-effectiveness analysis (CEA) | from enrollment to end of treatment at 12 months
  Incremental cost-effectiveness ratios (ICERs) will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Camaro, MD, Principal Investigator — Radboudumc / department Cardiology 616
Locations (1):
- Radboudumc Nijmegen, The Netherlands, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
It is anticipated that individual participant data (IPD) will be made available. A detailed and comprehensive data sharing strategy will be established in 2026

REFERENCES:
- See also: Related Info — https://projecten.zonmw.nl/nl/project/pehospitale-triage-van-patienten-met-intermediair-en-hoog-risico-op-acs-de-artica-2-trial